CLINICAL TRIAL: NCT06168292
Title: Intraductal Radiofrequency Thermoablation and Radiotherapy Combined Treatment for Extrahepatic Cholangiocarcinoma: A Prospective, Single-arm, Multicenter Study
Brief Title: Intraductal Radiofrequency Thermoablation and Radiotherapy Combined Treatment for Extrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Sang Myung Woo, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2023-0200
Record Dates: First submitted 2023-11-26; First posted 2023-12-13 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Biliary Tract Carcinoma; Radiotherapy; Radio-frequency Ablation
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): The clinical study will be conducted in the following order. Of patients with extrahepatic cholangiocarcinoma requiring biliary drainage, those who meet the inclusion criteria and consent to the study will be enrolled in the study and hospitalized to undergo endoscopic biliary drainage. The histologic or cytologic examination will be performed at the time of the first biliary drainage, and the extent of the cholangiocarcinoma lesion will be assessed during the procedure. After the diagnosis of extrahepatic cholangiocarcinoma, ID-RFA will be performed, and a biliary stent will be inserted for biliary drainage. Radiotherapy will be performed within 1 month of ID-RFA.
  Interventions: Procedure: ID-RFA and Radiotherapy

INTERVENTIONS:
Procedure: ID-RFA and Radiotherapy — The histologic or cytologic examination will be performed at the time of the first biliary drainage, and the extent of the cholangiocarcinoma lesion will be assessed during the procedure. After the diagnosis of extrahepatic cholangiocarcinoma, ID-RFA will be performed, and a biliary stent will be inserted for biliary drainage. Radiotherapy will be performed within 1 month of ID-RFA.

SUMMARY:
[Study objectives] To evaluate the efficacy and safety of the combined treatment of radiotherapy and endoscopic intraductal radiofrequency ablation in patients with locoregional extrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
○ Study flow The clinical study will be conducted in the following order. Of patients with extrahepatic cholangiocarcinoma requiring biliary drainage, those who meet the inclusion criteria and consent to the study will be enrolled in the study and hospitalized to undergo endoscopic biliary drainage. The histologic or cytologic examination will be performed at the time of the first biliary drainage, and the extent of the cholangiocarcinoma lesion will be assessed during the procedure. After the diagnosis of extrahepatic cholangiocarcinoma, ID-RFA will be performed, and a biliary stent will be inserted for biliary drainage. Radiotherapy will be performed within 1 month of ID-RFA.

Systemic chemotherapy is also one of the main treatments for patients with inoperable cholangiocarcinoma. Administration of subsequent chemotherapy is recommended after radiotherapy. The choice of chemotherapy regimen is at the discretion of the investigator based on on the patient's age, performance status, and other factors. For older patients who are inoperable, systemic chemotherapy may be difficult to administer.

Tumor response assessment will be performed using CT or MR every 2 months ± 2 weeks based on based on RECIST 1.1.

* Endoscopic biliary drainage The ERCP procedure is performed by an experienced pancreatobiliary endoscopist. A standardized endoscopic sphincterotomy (EST) is usually performed prior to stenting. If EST is difficult, a precut sphincterotomy may be performed first. After selective intubation into the bile duct according to the usual process of biliary drainage, a guidewire is placed upstream of the stricture and a biliary stent is inserted, and the type and length of the stent are selected at the discretion of the investigator. Systemic anti-cancer therapy after radiotherapy will be conducted at the discretion of the investigator, considering the patient's condition.
* ID-RFA ID-RFA requires a catheterized electrode that can be used through the channel of the ERCP. Currently, there are two commercially available RFA catheters: the Habib EndoHBP® (Boston Scientific, London, UK) and the ELRA RFA catheter® (Starmed, Goyang, Korea). This study uses the Habib catheter, which is an 8Fr bipolar catheter with two 8 mm electrodes that can be inserted into the bile duct by ERCP along a guidewire. The standard RFA is 7-10 W for 90 sec, and the energy and treatment time can be adjusted according to the operator's discretion. Repeated RFA can be performed by adjusting the catheter from proximal to distal depending on the length of the stricture during the same endoscopic session. After ID-RFA, a biliary stent is inserted to ensure bile duct patency and prevent stricture.
* Radiotherapy Radiotherapy is aimed to start within 1 month after ID-RFA. The radiotherapy dose will be 30-50 Gy in 10 fractions, considering the planning target volume based on the dose-volume standard.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 20 years of age or older, who voluntarily agree to participate in the study and sign the informed consent.
2. Patients with cytopathologically diagnosed inoperable extrahepatic cholangiocarcinoma

Exclusion Criteria:

1. Patients who refuse to sign the informed consent
2. Patients with metastatic cancer (stage IV) or malignant ascites
3. Patients with intrahepatic cholangiocarcinoma
4. Patients who are unable to undergo endoscopic procedures as determined by the investigator.
5. Patients with a life expectancy of 3 months or less
6. Patients with ID-RFA contraindications: pacemaker, pregnancy, uncorrected bleeding tendency (PT INR > 1.5, platelets < 50,000/mm3)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
2-year local control rate | At 2 years from the date of study enrollment
  2-year local control rate

SECONDARY OUTCOMES:
1-year local control rate | At 1 years from the date of study enrollment
  1-year local control rate
Overall survival | The time point of death from any cause from the study enrollment date, whichever occurs first, up to 2 years
  Overall survival
Progression-free survival | The time point of the date of study enrollment until disease progression or death from any cause, whichever occurs first, up to 2 years
  Progression-free survival
Local progression-free survival | The time point of the date of study enrollment until locoregional progression or death from any cause, whichever occurs first, up to 2 years
  Local progression-free survival
Period of Stent patency | The time point of the date of biliary stent placement after ID-RFA to the occurrence of stent dysfunction, up to 2 years
  Period of Stent patency

CONTACTS AND LOCATIONS:
Overall Officials: Sang Myung Woo, M.D, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Korea, Goyang-si, Other, South Korea

REFERENCES:
- [Background] Prezzano KM, Prasad D, Hermann GM, Belal AN, Alberico RA. Radiofrequency Ablation and Radiation Therapy Improve Local Control in Spinal Metastases Compared to Radiofrequency Ablation Alone. Am J Hosp Palliat Care. 2019 May;36(5):417-422. doi: 10.1177/1049909118819460. Epub 2018 Dec 13. PMID 30541334
- [Background] Hiraki T, Gobara H, Iguchi T, Fujiwara H, Matsui Y, Kanazawa S. Radiofrequency ablation for early-stage nonsmall cell lung cancer. Biomed Res Int. 2014;2014:152087. doi: 10.1155/2014/152087. Epub 2014 Jun 3. PMID 24995270
- [Background] Autorino R, Mattiucci GC, Ardito F, Balducci M, Deodato F, Macchia G, Mantini G, Perri V, Tringali A, Gambacorta MA, Tagliaferri L, Giuliante F, Morganti AG, Valentini V. Radiochemotherapy with Gemcitabine in Unresectable Extrahepatic Cholangiocarcinoma: Long-term Results of a Phase II Study. Anticancer Res. 2016 Feb;36(2):737-40. PMID 26851032
- [Background] Cho JH, Jeong S, Kim EJ, Kim JM, Kim YS, Lee DH. Long-term results of temperature-controlled endobiliary radiofrequency ablation in a normal swine model. Gastrointest Endosc. 2018 Apr;87(4):1147-1150. doi: 10.1016/j.gie.2017.09.013. Epub 2017 Sep 25. PMID 28958907
- [Background] Kim EJ, Chung DH, Kim YJ, Kim YS, Park YH, Kim KK, Cho JH. Endobiliary radiofrequency ablation for distal extrahepatic cholangiocarcinoma: A clinicopathological study. PLoS One. 2018 Nov 15;13(11):e0206694. doi: 10.1371/journal.pone.0206694. eCollection 2018. PMID 30439965
- [Background] Sofi AA, Khan MA, Das A, Sachdev M, Khuder S, Nawras A, Lee W. Radiofrequency ablation combined with biliary stent placement versus stent placement alone for malignant biliary strictures: a systematic review and meta-analysis. Gastrointest Endosc. 2018 Apr;87(4):944-951.e1. doi: 10.1016/j.gie.2017.10.029. Epub 2017 Nov 3. PMID 29108980
- [Background] Yang J, Wang J, Zhou H, Zhou Y, Wang Y, Jin H, Lou Q, Zhang X. Efficacy and safety of endoscopic radiofrequency ablation for unresectable extrahepatic cholangiocarcinoma: a randomized trial. Endoscopy. 2018 Aug;50(8):751-760. doi: 10.1055/s-0043-124870. Epub 2018 Jan 17. PMID 29342492
- [Background] Lee YN, Jeong S, Choi HJ, Cho JH, Cheon YK, Park SW, Kim YS, Lee DH, Moon JH. The safety of newly developed automatic temperature-controlled endobiliary radiofrequency ablation system for malignant biliary strictures: A prospective multicenter study. J Gastroenterol Hepatol. 2019 Aug;34(8):1454-1459. doi: 10.1111/jgh.14657. Epub 2019 Apr 14. PMID 30861593
- [Background] Klement RJ, Abbasi-Senger N, Adebahr S, Alheid H, Allgaeuer M, Becker G, Blanck O, Boda-Heggemann J, Brunner T, Duma M, Eble MJ, Ernst I, Gerum S, Habermehl D, Hass P, Henkenberens C, Hildebrandt G, Imhoff D, Kahl H, Klass ND, Krempien R, Lewitzki V, Lohaus F, Ostheimer C, Papachristofilou A, Petersen C, Rieber J, Schneider T, Schrade E, Semrau R, Wachter S, Wittig A, Guckenberger M, Andratschke N. The impact of local control on overall survival after stereotactic body radiotherapy for liver and lung metastases from colorectal cancer: a combined analysis of 388 patients with 500 metastases. BMC Cancer. 2019 Feb 26;19(1):173. doi: 10.1186/s12885-019-5362-5. PMID 30808323
- [Background] Machtay M, Paulus R, Moughan J, Komaki R, Bradley JE, Choy H, Albain K, Movsas B, Sause WT, Curran WJ. Defining local-regional control and its importance in locally advanced non-small cell lung carcinoma. J Thorac Oncol. 2012 Apr;7(4):716-22. doi: 10.1097/JTO.0b013e3182429682. PMID 22425920
- [Background] Gkika E, Hawkins MA, Grosu AL, Brunner TB. The Evolving Role of Radiation Therapy in the Treatment of Biliary Tract Cancer. Front Oncol. 2020 Dec 14;10:604387. doi: 10.3389/fonc.2020.604387. eCollection 2020. PMID 33381458
- [Background] Park N, Jung MK, Kim EJ, Paik WH, Cho JH. In-stent radiofrequency ablation with uncovered metal stent placement for tumor ingrowth/overgrowth causing self-expandable metal stent occlusion in distal malignant biliary obstruction: multicenter propensity score-matched study. Gastrointest Endosc. 2023 Apr;97(4):694-703.e2. doi: 10.1016/j.gie.2022.11.017. Epub 2022 Nov 30. PMID 36460085